CLINICAL TRIAL: NCT05419505
Title: APHRODITE-1: A Phase 2, Open Label, Self-Controlled Study of Different Interventions to Reduce Bruising Following CCH-Aaes Treatment for Cellulite of the Buttocks in Adult Females
Brief Title: Study of Different Interventions to Reduce Bruising Following CCH-Aaes Treatment for Cellulite of the Buttocks
Acronym: APHRODITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-226
Record Dates: First submitted 2022-06-09; First posted 2022-06-15 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Edematous Fibrosclerotic Panniculopathy; Cellulite
Keywords: Collagenase Clostridium Histolyticum; collagenase clostridium histolyticum-aaes
MeSH Terms: conditions — Cellulite | interventions — Antifibrinolytic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: CCH-aaes Dose Evaluation (Experimental): Participants will be administered CCH-aaes at different doses. Participants will receive CCH-aaes treatments in a split buttock arrangement, with the right buttock as the control, and the left buttock as the investigational treatment.
  Interventions: Drug: CCH-aaes
- Cohort 2: CCH-aaes Concentration Evaluation (Experimental): Participants will be administered CCH-aaes at different concentrations. Participants will receive CCH-aaes treatments in a split buttock arrangement, with the right buttock as the control, and the left buttock as the investigational treatment.
  Interventions: Drug: CCH-aaes
- Cohort 3: CCH-aaes Injection Depth Evaluation (Experimental): Participants will be administered CCH-aaes using different injection depths. Participants will receive CCH-aaes treatments in a split buttock arrangement, with the right buttock as the control, and the left buttock as the investigational treatment.
  Interventions: Drug: CCH-aaes
- Cohort 4: CCH-aaes Injection Method Evaluation (Experimental): Participants will be administered CCH-aaes using different injection methods. Participants will receive CCH-aaes treatments in a split buttock arrangement, with the right buttock as the control, and the left buttock as the investigational treatment.
  Interventions: Drug: CCH-aaes
- Cohort 5: CCH-aaes and Diluent Additive Evaluation (Experimental): Participants will be administered CCH-aaes and diluent additive. Participants will receive CCH-aaes treatments in a split buttock arrangement, with the right buttock as the control, and the left buttock as the investigational treatment.
  Interventions: Drug: CCH-aaes
- Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation (Experimental): Participants will be administered CCH-aaes using a different treatment schedule and different doses and concentrations. Participants will receive CCH-aaes treatments in a split buttock arrangement, with the right buttock as the control, and the left buttock as the investigational treatment.
  Interventions: Drug: CCH-aaes
- Cohort 7: CCH-aaes and Antifibrinolytic Agent (Experimental): Participants will be administered CCH-aaes and an antifibrinolytic agent. Participants will receive CCH-aaes treatments in a split buttock arrangement, with the right buttock as the control, and the left buttock as the investigational treatment.
  Interventions: Drug: CCH-aaes; Drug: Antifibrinolytic Agent

INTERVENTIONS:
Drug: CCH-aaes — Administered by subcutaneous injection.
  Other Names: Collagenase clostridium histolyticum-aaes; QWO®
Drug: Antifibrinolytic Agent — Self-administered by participants enrolled in Cohort 7.
  Arms: Cohort 7: CCH-aaes and Antifibrinolytic Agent

SUMMARY:
The study will evaluate the effect of different doses, strengths (concentrations), diluent additives, depths of injection, and methods of injection on the severity of bruising potentially induced by QWO (collagenase clostridium histolyticum-aaes [CCH-aaes]).

DETAILED DESCRIPTION:
The study will comprise a Screening Period (28 days), Treatment Period (90 days), and Follow-up Period (90 days). Participants will receive CCH-aaes in different doses, concentrations, diluent additives, depths of injection, and methods of injection in a split buttock arrangement, with the right buttock serving as the control, and the left buttock (investigational side) receiving a study intervention.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index of 18 to <32 kilograms (kg)/meter (m)^2 and intends to maintain stable body weight during the study.
* Have both buttocks with moderate or severe cellulite as reported by the investigator using the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS).
* Have a Hexsel Cellulite Severity Scale (CSS) Total Score of ≤12.
* Has a Fitzpatrick Skin Type of I-IV
* Be willing to apply sunscreen to the treatment areas before each exposure to the sun for the duration of participation in the study.
* Be willing and able to comply with the requirements of the study.

Key Exclusion Criteria:

* Has systemic conditions (coagulation disorders, skin pigmentation disorders, malignancy, keloidal scarring, abnormal wound healing) that restricts study participation.
* Is pregnant and/or is breast-feeding or plans to become pregnant and/or to breast-feed during the course of the study.
* Has any local (in the areas to be treated) conditions (thrombosis, post-thrombosis syndrome, vascular disorder, inflammation, active infection, active cutaneous alteration, tattoo or mole) that restricts study participation.
* Requires antiplatelet medication, anticoagulants, or non-steroidal anti-inflammatory drugs during the study.
* Any medications, supplements, or foods that have, or have been reported to have anticoagulant effects within 14 days of treatment.
* Has received treatment with investigational treatment within 30 days before treatment.
* Has used or intends to use any of the local applications, therapies, injections, or procedures for the treatment of cellulite on either buttock that would restrict study participation.
* Intends to initiate an intensive sport or exercise program or intensive weight reduction program during the study.
* Intends to engage in strenuous activity within 48 hours of study intervention administration.
* Has recently tanned or intends to tan (outdoors or indoors) during the study.
* Has a history of hypersensitivity or allergy to collagenase or any other excipient of CCH.
* Has any condition(s) that, in the investigator's opinion, might indicate the participant to be unsuitable for the study.
* Has participated in a previous investigational study of CCH or received any collagenase treatments at any time prior to treatment in this study for the treatment of cellulite of the buttocks.

In addition to the applicable aforementioned exclusion criteria, participants enrolling in Cohort 7 will be excluded from study participation if the participant:

* Has any of the following medical conditions:

  1. history of venous or arterial thromboembolism or current thromboembolic disease.
  2. history of or current renal impairment.
  3. serum creatinine concentration > 1.4 milligram/deciliter at Screening.
* Requires the following concomitant medications during the study and cannot discontinue these medications within the time specified before CCH-aaes treatment:

  1. concurrently taking combination hormonal contraceptives.
  2. concurrently undergoing hormone replacement therapy.
  3. is a current smoker of nicotine or cannabinoids.
* Participants in Cohort 7 should avoid smoking (including vaping, nicotine, or marijuana cigarettes) during the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hernandez, Study Director — Endo Pharmaceuticals
Locations (13):
- United States (13):
  - Endo Clinical Trial Site #6, Scottsdale, Arizona
  - Endo Clinical Trial Site #4, Beverly Hills, California
  - Endo Clinical Trial Site #9, Encinitas, California
  - Endo Clinical Trial Site #10, San Diego, California
  - Endo Clinical Trial Site #7, Solana Beach, California
  - Endo Clinical Trial Site #12, Greenwood Village, Colorado
  - Endo Clinical Trial Site #8, Coral Gables, Florida
  - Endo Clinical Trial Site #13, Miami, Florida
  - Endo Clinical Trial Site #3, Chicago, Illinois
  - Endo Clinical Trial Site #2, Metairie, Louisiana
  - Endo Clinical Trial Site #11, New York, New York
  - Endo Clinical Trial Site #1, Nashville, Tennessee
  - Endo Clinical Trial Site #5, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety-one participants were enrolled in this split-person study to compare different collagenase clostridium histolyticum-aaes (CCH-aaes) treatment regimens. Participants were administered study intervention in a split-buttock arrangement, with each participant's right buttock serving as the control to their assigned intervention administered to the left buttock (test).
Units Other Than Participants: buttock
Groups:
- Cohort 1: CCH-aaes Dose Evaluation: Test: Participants left buttock (test) received CCH-aaes injection using half the labeled dose (0.42 milligrams [mg]) but maintaining the labeled concentration (0.23 mg/milliliters [mL]).
  Control: Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
- Cohort 2: CCH-aaes Concentration Evaluation: Test: Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) but using an approximate 5-fold dilution (0.05 mg/mL) of the labeled concentration (0.23 mg/mL).
  Control: Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
- Cohort 3: CCH-aaes Injection Depth Evaluation: Test: Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) but with an injection depth of one-quarter inch.
  Control: Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) with labeled injection depth of one-half inch.
- Cohort 4: CCH-aaes Injection Method Evaluation: Test: Participants left buttock (test) received CCH-aaes injection using an approximate 2.5-fold dilution of the labeled concentration (0.09 mg/mL) but administering only a single aliquot at one-quarter-inch depth per injection administered at up to 30 injections.
  Control" Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) but administering only a single aliquot at one-quarter-inch depth per injection administered at up to 12 injections.
- Cohort 5: CCH-aaes and Diluent Additive Evaluation: Test: Participants left buttock (test) received CCH-aaes injection using half the labeled dose (0.42 mg) with diluent additive.
  Control: Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
- Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation: Test: Participants left buttock (test) received CCH-aaes injection using one-quarter of the labeled dose (0.21 mg) at one-half the labeled concentration (0.12 mg/mL). Treatment sessions were administered 6 weeks apart.
  Control: Participants right buttock (control) received CCH-aaes injection using one-half the labeled dose (0.42 mg) but maintaining the labeled concentration (0.23 mg/mL). Treatment sessions were administered 6 weeks apart.
- Cohort 7a: CCH-aaes and Antifibrinolytic Agent; Cohort 7b: CCH-aaes and Antifibrinolytic Agent: Test: Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) with an antifibrinolytic agent treatment regimen.
  Control: Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
Period: Overall Study
Arm/Group | Cohort 1: CCH-aaes Dose Evaluation | Cohort 2: CCH-aaes Concentration Evaluation | Cohort 3: CCH-aaes Injection Depth Evaluation | Cohort 4: CCH-aaes Injection Method Evaluation | Cohort 5: CCH-aaes and Diluent Additive Evaluation | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation | Cohort 7a: CCH-aaes and Antifibrinolytic Agent | Cohort 7b: CCH-aaes and Antifibrinolytic Agent
Started | 22; 44 buttock (Left and right buttock) | 14; 28 buttock (Left and right buttock) | 5; 10 buttock (Left and right buttock) | 7; 14 buttock (Left and right buttock) | 10; 20 buttock (Left and right buttock) | 19; 38 buttock (Left and right buttock) | 7; 14 buttock (Left and right buttock) | 7; 14 buttock (Left and right buttock)
Completed | 19; 38 buttock | 11; 22 buttock | 5; 10 buttock | 6; 12 buttock | 9; 18 buttock | 17; 34 buttock | 6; 12 buttock | 6; 12 buttock
Not Completed | 3; 6 buttock | 3; 6 buttock | 0; 0 buttock | 1; 2 buttock | 1; 2 buttock | 2; 4 buttock | 1; 2 buttock | 1; 2 buttock
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 injection of CCH-aaes.
Groups:
- Cohort 1: CCH-aaes Dose Evaluation: Participants left buttock (test) received CCH-aaes injection using half the labeled dose (0.42 milligrams [mg]) but maintaining the labeled concentration (0.23 mg/milliliters [mL]).
  Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL)
- Cohort 2: CCH-aaes Concentration Evaluation: Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) but using an approximate 5-fold dilution (0.05 mg/mL) of the labeled concentration (0.23 mg/mL).
  Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
- Cohort 3: CCH-aaes Injection Depth Evaluation: Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) but with an injection depth of one-quarter inch.
  Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) with labeled injection depth of one-half inch.
- Cohort 4: CCH-aaes Injection Method Evaluation: Participants left buttock (test) received CCH-aaes injection using an approximate 2.5-fold dilution of the labeled concentration (0.09 mg/mL) but administering only a single aliquot at one-quarter-inch depth per injection administered at up to 30 injections.
  Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) but administering only a single aliquot at one-quarter-inch depth per injection administered at up to 12 injections.
- Cohort 5: CCH-aaes and Diluent Additive Evaluation: Participants left buttock (test) received CCH-aaes injection using half the labeled dose (0.42 mg) with diluent additive.
  Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
- Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation: Participants left buttock (test) received CCH-aaes injection using one-quarter of the labeled dose (0.21 mg) at one-half the labeled concentration (0.12 mg/mL). Treatment sessions were administered 6 weeks apart.
  Participants right buttock (control) received CCH-aaes injection using one-half the labeled dose (0.42 mg) but maintaining the labeled concentration (0.23 mg/mL). Treatment sessions were administered 6 weeks apart.
- Cohort 7a: CCH-aaes and Antifibrinolytic Agent; Cohort 7b: CCH-aaes and Antifibrinolytic Agent: Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) with an antifibrinolytic agent treatment regimen.
  Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: CCH-aaes Dose Evaluation | Cohort 2: CCH-aaes Concentration Evaluation | Cohort 3: CCH-aaes Injection Depth Evaluation | Cohort 4: CCH-aaes Injection Method Evaluation | Cohort 5: CCH-aaes and Diluent Additive Evaluation | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation | Cohort 7a: CCH-aaes and Antifibrinolytic Agent | Cohort 7b: CCH-aaes and Antifibrinolytic Agent | Total
Number analyzed (Participants) | 22 | 14 | 5 | 7 | 10 | 19 | 7 | 7 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.50 (10.698) | 44.79 (9.125) | 44.40 (8.503) | 34.00 (8.699) | 46.50 (10.179) | 47.74 (7.225) | 37.57 (10.967) | 38.57 (10.549) | 43.40 (9.998)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 14 | 5 | 7 | 10 | 19 | 7 | 7 | 91
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 18 | 14 | 5 | 7 | 9 | 18 | 6 | 7 | 84
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Multiple | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1-Level Lower Score 3 to 5 Days After Initial CCH-aaes Injection, as Assessed by the Investigator Assessment of Bruising Severity Scale (IABSS) After Initial CCH-aaes Injection
Description: The investigator assessed the severity of bruising using the IABSS, The IABSS is a 5-point scale ranging from 0-4, with 0 indicating no bruising or almost none, and 4 indicating very severe bruising. Higher scores indicated worse outcomes.
  The investigator compared the bruising of the left (test) buttock to the right (control) buttock. Responders were participants whose left buttock/test side demonstrated at least a 1-level lower IABSS score versus the right buttock/control side.
  Percentages are based on the number of participants with an assessment at specified timepoint.
Time Frame: 3 to 5 days after initial CCH-aaes injection of left buttock (test) and right buttock (control)
Population: All participants who received at least 1 injection of CCH-aaes and who had at least 1 valid IABSS assessment after an injection of CCH-aaes at specified timepoint. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: CCH-aaes Dose Evaluation | Cohort 2: CCH-aaes Concentration Evaluation | Cohort 3: CCH-aaes Injection Depth Evaluation | Cohort 4: CCH-aaes Injection Method Evaluation | Cohort 5: CCH-aaes and Diluent Additive Evaluation | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation | Cohort 7a: CCH-aaes and Antifibrinolytic Agent | Cohort 7b: CCH-aaes and Antifibrinolytic Agent
Number analyzed (Participants) | 21 | 12 | 5 | 6 | 9 | 19 | 6 | 6
percentage of participants | 90.5 [69.62 to 98.83] | 25.0 [5.49 to 57.19] | 20.0 [0.51 to 71.64] | 33.3 [4.33 to 77.72] | 44.4 [13.70 to 78.80] | 63.2 [38.36 to 83.71] | 33.3 [4.33 to 77.72] | 33.3 [4.33 to 77.72]

2. Secondary Outcome: Percentage of Participants With at Least 1-Level Lower Score, as Assessed by the IABSS
Description: The investigator assessed the severity of bruising using the IABSS, The IABSS is a 5-point scale ranging from 0-4, with 0 indicating no bruising or almost none, and 4 indicating very severe bruising. Higher scores indicated worse outcome.
  The investigator compared the bruising of the left buttock (test) to the right (control) buttock. Responders were participants whose left buttock/test side at Visit A demonstrated at least a 1-level lower IABSS score versus the right buttock/control side at Visit B, where Visit A and B could either be the same or different. Follow-up after first injection is presented: Follow-up 1 is 1 to 2 days after injection visit, Follow-up 2 is 3 to 5 days after injection visit, Follow-up 3 is 6 to 9 days after injection visit, and Follow-up 4 is 10 to 14 days after injection visit.
  Percentages are based on the number of participants with an assessment at specified timepoint.
Time Frame: Follow-up 1, 2, 3, and 4 after CCH-aaes injection of left buttock (test) and right buttock (control)
Population: All participants who received at least 1 injection of CCH-aaes and who had at least 1 valid IABSS assessment after an injection of CCH-aaes at specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1: CCH-aaes Dose Evaluation: Participants left buttock (test) received CCH-aaes injection using half the labeled dose (0.42 mg) but maintaining the labeled concentration (0.23 mg/mL).
  Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
Arm/Group | Cohort 1: CCH-aaes Dose Evaluation | Cohort 2: CCH-aaes Concentration Evaluation | Cohort 3: CCH-aaes Injection Depth Evaluation | Cohort 4: CCH-aaes Injection Method Evaluation | Cohort 5: CCH-aaes and Diluent Additive Evaluation | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation | Cohort 7a: CCH-aaes and Antifibrinolytic Agent | Cohort 7b: CCH-aaes and Antifibrinolytic Agent
Number analyzed (Participants) | 22 | 14 | 5 | 7 | 10 | 19 | 7 | 7
percentage of participants
  Follow-up 1: number analyzed (Participants) | 22 | 13 | 5 | 7 | 10 | 18 | 6 | 7
  Follow-up 1 | 81.8 [59.72 to 94.81] | 15.4 [1.92 to 45.45] | 0 [0 to 52.18] | 42.9 [9.90 to 81.59] | 40.0 [12.16 to 73.76] | 44.4 [21.53 to 69.24] | 16.7 [0.42 to 64.12] | 42.9 [9.90 to 81.59]
  Follow-up 2: number analyzed (Participants) | 21 | 12 | 5 | 6 | 9 | 19 | 6 | 6
  Follow-up 2 | 90.5 [69.62 to 98.83] | 25.0 [5.49 to 57.19] | 20.0 [0.51 to 71.64] | 33.3 [4.33 to 77.72] | 44.4 [13.70 to 78.80] | 63.2 [38.36 to 83.71] | 33.3 [4.33 to 77.72] | 33.3 [4.33 to 77.72]
  Follow-up 3: number analyzed (Participants) | 22 | 13 | 5 | 7 | 10 | 19 | 5 | 7
  Follow-up 3 | 40.9 [20.71 to 63.65] | 38.5 [13.86 to 68.42] | 40.0 [5.27 to 85.34] | 28.6 [3.67 to 70.96] | 10.0 [0.25 to 44.50] | 31.6 [12.58 to 56.55] | 40.0 [5.27 to 85.34] | 42.9 [9.90 to 81.59]
  Follow-up 4: number analyzed (Participants) | 22 | 11 | 5 | 7 | 10 | 19 | 6 | 7
  Follow-up 4 | 13.6 [2.91 to 34.91] | 18.2 [2.28 to 51.78] | 0 [0 to 52.18] | 14.3 [0.36 to 57.87] | 10.0 [0.25 to 44.50] | 21.1 [6.05 to 45.57] | 16.7 [0.42 to 64.12] | 71.4 [29.04 to 96.33]

3. Secondary Outcome: Percentage of Participants With at Least +1 or Higher Score on the Investigator-Global Aesthetic Improvement Scale (I-GAIS) After CCH-aaes Injection
Description: The investigator determined the degree of improvement of each buttock by comparing treated cellulite dimples from the Day 1 pre-treatment (Baseline) digital image of each buttock to the treated dimples observed in a live assessment.
  The investigator determined the degree of improvement of each buttock with the I-GAIS, which uses a 7-point scale ranging from +3 (very much improved) to -3 (very much worse). A higher score indicated a better outcome. The investigator compared the bruising of the left (test) buttock to the right (control) buttock.
  A 1-level I-GAIS responder was defined as any participant with an improved (+1, +2 or +3) score on the I-GAIS at an analysis visit for that treatment area.
  Percentages are based on the number of participants with an assessment at specified timepoint.
Time Frame: Day 22 and Day 43 for Cohorts 1 to 5, Day 43 for Cohort 6, Day 22, Day 43, and Day 64 for Cohort 7, and Day 90, Day 135, and Day 180 for all cohorts
Population: All participants who received at least 1 injection of CCH-aaes and who had at least 1 valid assessment at a treatment area after an injection of CCH-aaes.
  For Cohort 7a, on Day 22, I-GAIS was only assessed for the investigational buttock (left buttock) and for Cohort 7b, on Day 22, I-GAIS was only assessed for the control buttock (right buttock).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: CCH-aaes Dose Evaluation | Cohort 2: CCH-aaes Concentration Evaluation | Cohort 3: CCH-aaes Injection Depth Evaluation | Cohort 4: CCH-aaes Injection Method Evaluation | Cohort 5: CCH-aaes and Diluent Additive Evaluation | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation | Cohort 7a: CCH-aaes and Antifibrinolytic Agent | Cohort 7b: CCH-aaes and Antifibrinolytic Agent
Number analyzed (Participants) | 21 | 13 | 5 | 6 | 10 | 18 | 7 | 7
percentage of participants
  Day 22 Left Buttock (Test): number analyzed (Participants) | 21 | 12 | 5 | 6 | 10 | 0 | 7 | 0
  Day 22 Left Buttock (Test) | 42.9 [21.82 to 65.98] | 58.3 [27.67 to 84.83] | 100 [47.82 to 100] | 66.7 [22.28 to 95.67] | 40.0 [12.16 to 73.76] |  | 85.7 [42.13 to 99.64] |
  Day 22 Right Buttock (Control): number analyzed (Participants) | 21 | 12 | 5 | 6 | 10 | 0 | 0 | 7
  Day 22 Right Buttock (Control) | 57.1 [34.02 to 78.18] | 66.7 [34.89 to 90.08] | 100 [47.82 to 100] | 66.7 [22.28 to 95.67] | 40.0 [12.16 to 73.76] |  |  | 100 [59.04 to 100]
  Day 43 Left Buttock (Test): number analyzed (Participants) | 21 | 13 | 5 | 6 | 9 | 18 | 5 | 7
  Day 43 Left Buttock (Test) | 71.4 [47.82 to 88.72] | 84.6 [54.55 to 98.08] | 100 [47.82 to 100] | 83.3 [35.88 to 99.58] | 66.7 [29.93 to 92.51] | 44.4 [21.53 to 69.24] | 100 [47.82 to 100] | 100 [59.04 to 100]
  Day 43 Right Buttock (Control): number analyzed (Participants) | 21 | 13 | 5 | 6 | 9 | 18 | 5 | 7
  Day 43 Right Buttock (Control) | 76.2 [52.83 to 91.78] | 76.9 [46.19 to 94.96] | 100 [47.82 to 100] | 100 [54.07 to 100] | 66.7 [29.93 to 92.51] | 50.0 [26.02 to 73.98] | 40.0 [5.27 to 85.34] | 100 [59.94 to 100]
  Day 64 Left Buttock (Test): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7
  Day 64 Left Buttock (Test) |  |  |  |  |  |  | 100 [47.82 to 100] | 100 [59.04 to 100]
  Day 64 Right Buttock (Control): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7
  Day 64 Right Buttock (Control) |  |  |  |  |  |  | 100 [47.82 to 100] | 100 [59.04 to 100]
  Day 90 (Follow-up) Left Buttock (Test): number analyzed (Participants) | 21 | 10 | 5 | 6 | 9 | 18 | 7 | 7
  Day 90 (Follow-up) Left Buttock (Test) | 38.1 [18.11 to 61.56] | 70.0 [34.75 to 93.33] | 100 [47.82 to 100] | 66.7 [22.8 to 95.67] | 44.4 [13.70 to 78.80] | 27.8 [9.69 to 53.48] | 85.7 [42.13 to 99.64] | 100 [59.04 to 100]
  Day 90 (Follow-up) Right Buttock (Control): number analyzed (Participants) | 21 | 10 | 5 | 6 | 9 | 18 | 7 | 7
  Day 90 (Follow-up) Right Buttock (Control) | 47.6 [25.71 to 70.22] | 80.0 [44.39 to 97.48] | 100 [47.82 to 100] | 83.3 [35.88 to 99.58] | 44.4 [13.70 to 78.80] | 38.9 [17.30 to 64.25] | 71.4 [29.04 to 96.33] | 100 [59.04 to 100]
  Day 135 (Follow-up) Left Buttock (Test): number analyzed (Participants) | 19 | 11 | 5 | 6 | 9 | 18 | 6 | 6
  Day 135 (Follow-up) Left Buttock (Test) | 36.8 [16.29 to 61.64] | 90.9 [58.72 to 99.77] | 100 [47.82 to 100] | 50.0 [11.81 to 88.19] | 22.2 [2.81 to 60.01] | 22.2 [6.41 to 47.64] | 83.3 [35.88 to 99.58] | 100 [54.07 to 100]
  Day 135 (Follow-up) Right Buttock (Control): number analyzed (Participants) | 19 | 11 | 5 | 6 | 9 | 18 | 6 | 6
  Day 135 (Follow-up) Right Buttock (Control) | 47.4 [24.45 to 71.14] | 81.8 [48.22 to 97.72] | 100 [47.82 to 100] | 66.7 [22.28 to 95.67] | 22.2 [2.81 to 60.01] | 33.3 [13.34 to 59.01] | 66.7 [22.28 to 95.67] | 83.3 [35.88 to 99.58]
  Day 180 (End of Study) Left Buttock (Test): number analyzed (Participants) | 19 | 11 | 5 | 6 | 9 | 17 | 6 | 6
  Day 180 (End of Study) Left Buttock (Test) | 36.8 [16.29 to 61.64] | 100 [71.51 to 100] | 100 [47.82 to 100] | 50.0 [11.81 to 88.19] | 11.1 [0.28 to 48.25] | 17.6 [3.80 to 43.43] | 66.7 [22.28 to 95.67] | 83.3 [35.88 to 99.58]
  Day 180 (End of Study) Right Buttock (Control): number analyzed (Participants) | 19 | 11 | 5 | 6 | 9 | 17 | 6 | 6
  Day 180 (End of Study) Right Buttock (Control) | 36.8 [16.29 to 61.64] | 81.8 [48.22 to 97.72] | 100 [47.82 to 100] | 66.7 [22.28 to 95.67] | 11.1 [0.28 to 48.25] | 41.2 [18.44 to 67.08] | 66.7 [22.28 to 95.67] | 83.3 [35.88 to 99.58]

4. Secondary Outcome: Percentage of Participants With Injection Site Reactions
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse events (AEs) that occur or worsen (increase in severity) on the same day or after the study intervention administration on Day 1. Percent of participants with TEAEs of injection site reactions are presented by left buttock (test) and right buttock (control).
  A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From Day 1 (after dose) through Day 180
Population: All participants who received at least 1 injection of CCH-aaes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: CCH-aaes Dose Evaluation | Cohort 2: CCH-aaes Concentration Evaluation | Cohort 3: CCH-aaes Injection Depth Evaluation | Cohort 4: CCH-aaes Injection Method Evaluation | Cohort 5: CCH-aaes and Diluent Additive Evaluation | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation | Cohort 7a: CCH-aaes and Antifibrinolytic Agent | Cohort 7b: CCH-aaes and Antifibrinolytic Agent
Number analyzed (Participants) | 22 | 14 | 5 | 7 | 10 | 19 | 7 | 7
percentage of participants
  Left Buttock (Test) | 100 [84.56 to 100] | 92.9 [75.29 to 100] | 100 [47.82 to 100] | 100 [59.04 to 100] | 100 [69.15 to 100] | 100 [82.35 to 100] | 100 [59.04 to 100] | 100 [59.04 to 100]
  Right Buttock (Control) | 100 [84.56 to 100] | 92.9 [75.29 to 100] | 100 [47.82 to 100] | 100 [59.04 to 100] | 100 [69.15 to 100] | 100 [82.35 to 100] | 85.7 [54.07 to 100] | 100 [59.04 to 100]

ADVERSE EVENTS:
Time Frame: From Day 1 (after dose) through Day 180
Description: Data on all-cause mortality and serious adverse events were collected irrespective of the event's relation to the buttocks (test/control). The buttock Arms were limited to the analysis of localized events of the injection site region (ISR) only.
Groups:
- Cohort 1: CCH-aaes Dose Evaluation-Test (ISR): Participants left buttock (test) received CCH-aaes injection using half the labeled dose (0.42 mg) but maintaining the labeled concentration (0.23 mL).
- Cohort 1: CCH-aaes Dose Evaluation-Control (ISR); Cohort 2: CCH-aaes Concentration Evaluation -Control (ISR); Cohort 5: CCH-aaes and Diluent Additive Evaluation-Control (ISR); Cohort 7a: CCH-aaes and Antifibrinolytic Agent-Control (ISR); Cohort 7b: CCH-aaes and Antifibrinolytic Agent-Control (ISR): Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL).
- Cohort 2: CCH-aaes Concentration Evaluation-Test (ISR): Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) but using an approximate 5-fold dilution (0.05 mg/mL) of the labeled concentration (0.23 mg/mL).
- Cohort 3: CCH-aaes Injection Depth Evaluation-Test (ISR): Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) but with an injection depth of one-quarter inch.
- Cohort 3: CCH-aaes Injection Depth Evaluation-Control (ISR): Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) with labeled injection depth of one-half inch.
- Cohort 4: CCH-aaes Injection Method Evaluation-Test (ISR): Participants left buttock (test) received CCH-aaes injection using an approximate 2.5-fold dilution of the labeled concentration (0.09 mg/mL) but administering only a single aliquot at one-quarter-inch depth per injection administered at up to 30 injections.
- Cohort 4: CCH-aaes Injection Method Evaluation-Control (ISR): Participants right buttock (control) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) but administering only a single aliquot at one-quarter-inch depth per injection administered at up to 12 injections.
- Cohort 5: CCH-aaes and Diluent Additive Evaluation-Test (ISR): Participants left buttock (test) received CCH-aaes injection using half the labeled dose (0.42 mg) with diluent additive.
- Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation -Test (ISR): Participants left buttock (test) received CCH-aaes injection using one-quarter of the labeled dose (0.21 mg) at one-half the labeled concentration (0.12 mg/mL). Treatment sessions were administered 6 weeks apart.
- Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation-Control (ISR): Participants right buttock (control) received CCH-aaes injection using one-half the labeled dose (0.42 mg) but maintaining the labeled concentration (0.23 mg/mL). Treatment sessions were administered 6 weeks apart.
- Cohort 7a: CCH-aaes and Antifibrinolytic Agent-Test (ISR); Cohort 7b: CCH-aaes and Antifibrinolytic Agent-Test (ISR): Participants left buttock (test) received CCH-aaes injection using the labeled dose (0.84 mg) and concentration (0.23 mg/mL) with an antifibrinolytic agent treatment regimen.
- Cohort 1: Systemic/Non-ISR AEs: Adverse events that affected participants as a whole (systemic events) or non-injection site reactions in Cohort 1.
- Cohort 2: Systemic/Non-ISR AEs: Adverse events that affected participants as a whole (systemic events) or non-injection site reactions in Cohort 2.
- Cohort 3: Systemic/Non-ISR AEs: Adverse events that affected participants as a whole (systemic events) or non-injection site reactions in Cohort 3.
- Cohort 4: Systemic/Non-ISR AEs: Adverse events that affected participants as a whole (systemic events) or non-injection site reactions in Cohort 4.
- Cohort 5: Systemic/Non-ISR AEs: Adverse events that affected participants as a whole (systemic events) or non-injection site reactions in Cohort 5.
- Cohort 6: Systemic/Non-ISR AEs: Adverse events that affected participants as a whole (systemic events) or non-injection site reactions in Cohort 6.
- Cohort 7a: Systemic/Non-ISR AEs: Adverse events that affected participants as a whole (systemic events) or non-injection site reactions in Cohort 7a.
- Cohort 7b: Systemic/Non-ISR AEs: Adverse events that affected participants as a whole (systemic events) or non-injection site reactions in Cohort 7b.
Arm/Group | Cohort 1: CCH-aaes Dose Evaluation-Test (ISR) | Cohort 1: CCH-aaes Dose Evaluation-Control (ISR) | Cohort 2: CCH-aaes Concentration Evaluation-Test (ISR) | Cohort 2: CCH-aaes Concentration Evaluation -Control (ISR) | Cohort 3: CCH-aaes Injection Depth Evaluation-Test (ISR) | Cohort 3: CCH-aaes Injection Depth Evaluation-Control (ISR) | Cohort 4: CCH-aaes Injection Method Evaluation-Test (ISR) | Cohort 4: CCH-aaes Injection Method Evaluation-Control (ISR) | Cohort 5: CCH-aaes and Diluent Additive Evaluation-Test (ISR) | Cohort 5: CCH-aaes and Diluent Additive Evaluation-Control (ISR) | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation -Test (ISR) | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation-Control (ISR) | Cohort 7a: CCH-aaes and Antifibrinolytic Agent-Test (ISR) | Cohort 7a: CCH-aaes and Antifibrinolytic Agent-Control (ISR) | Cohort 7b: CCH-aaes and Antifibrinolytic Agent-Test (ISR) | Cohort 7b: CCH-aaes and Antifibrinolytic Agent-Control (ISR) | Cohort 1: Systemic/Non-ISR AEs | Cohort 2: Systemic/Non-ISR AEs | Cohort 3: Systemic/Non-ISR AEs | Cohort 4: Systemic/Non-ISR AEs | Cohort 5: Systemic/Non-ISR AEs | Cohort 6: Systemic/Non-ISR AEs | Cohort 7a: Systemic/Non-ISR AEs | Cohort 7b: Systemic/Non-ISR AEs
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/22 | 0/14 | 0/5 | 0/7 | 0/10 | 0/19 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/22 | 0/14 | 0/5 | 0/7 | 0/10 | 0/19 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22 | 13/14 | 13/14 | 5/5 | 5/5 | 7/7 | 7/7 | 10/10 | 10/10 | 19/19 | 19/19 | 7/7 | 6/7 | 7/7 | 7/7 | 4/22 | 0/14 | 3/5 | 0/7 | 0/10 | 4/19 | 0/7 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort 1: CCH-aaes Dose Evaluation-Test (ISR) (N=22) | Cohort 1: CCH-aaes Dose Evaluation-Control (ISR) (N=22) | Cohort 2: CCH-aaes Concentration Evaluation-Test (ISR) (N=14) | Cohort 2: CCH-aaes Concentration Evaluation -Control (ISR) (N=14) | Cohort 3: CCH-aaes Injection Depth Evaluation-Test (ISR) (N=5) | Cohort 3: CCH-aaes Injection Depth Evaluation-Control (ISR) (N=5) | Cohort 4: CCH-aaes Injection Method Evaluation-Test (ISR) (N=7) | Cohort 4: CCH-aaes Injection Method Evaluation-Control (ISR) (N=7) | Cohort 5: CCH-aaes and Diluent Additive Evaluation-Test (ISR) (N=10) | Cohort 5: CCH-aaes and Diluent Additive Evaluation-Control (ISR) (N=10) | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation -Test (ISR) (N=19) | Cohort 6: CCH-aaes Dose, Concentration, and Treatment Schedule Evaluation-Control (ISR) (N=19) | Cohort 7a: CCH-aaes and Antifibrinolytic Agent-Test (ISR) (N=7) | Cohort 7a: CCH-aaes and Antifibrinolytic Agent-Control (ISR) (N=7) | Cohort 7b: CCH-aaes and Antifibrinolytic Agent-Test (ISR) (N=7) | Cohort 7b: CCH-aaes and Antifibrinolytic Agent-Control (ISR) (N=7) | Cohort 1: Systemic/Non-ISR AEs (N=22) | Cohort 2: Systemic/Non-ISR AEs (N=14) | Cohort 3: Systemic/Non-ISR AEs (N=5) | Cohort 4: Systemic/Non-ISR AEs (N=7) | Cohort 5: Systemic/Non-ISR AEs (N=10) | Cohort 6: Systemic/Non-ISR AEs (N=19) | Cohort 7a: Systemic/Non-ISR AEs (N=7) | Cohort 7b: Systemic/Non-ISR AEs (N=7)
Injection site bruising (General disorders) | 22 | 22 | 13 | 13 | 5 | 5 | 0 | 0 | 10 | 10 | 19 | 19 | 0 | 0 | 7 | 7 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Injection site pain (General disorders) | 7 | 8 | 0 | 0 | 1 | 1 | 0 | 0 | 9 | 9 | 2 | 2 | 2 | 0 | 1 | 3 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Injection site discolouration (General disorders) | 10 | 10 | 0 | 0 | 3 | 3 | 2 | 2 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 0 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — All AEs classified as injection site hemorrhage (preferred MedDRA term) for reporting purposes were identified with the verbatim term "ecchymosis" by investigators during the study.
Injection site nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 2 | 2 | 1 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Injection site mass (General disorders) | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Injection site pruritus (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Injection site swelling (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Injection site papule (General disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Hypertension (Vascular disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was halted before the predetermined sample size was enrolled, therefore, was not adequately powered to draw conclusions or to make comparisons between cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT05419505/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT05419505/SAP_001.pdf